CLINICAL TRIAL: NCT01816204
Title: Therapist Assisted Online Treatment for Anxiety
Acronym: TAO-anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 539-2012
Record Dates: First submitted 2013-03-11; First posted 2013-03-22 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2015-04

CONDITIONS: Anxiety Disorders
Keywords: anxiety treatment; anxiety online treatment; anxiety electronic treatment; anxiety therapist assisted
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapist assisted online treatment (TAO) (Experimental): Students assigned to treatment with weekly online modules and weekly 10-15 minute video conference with counselor.
  Interventions: Behavioral: Therapist assisted online treatment
- face-to-face individual therapy (Active Comparator): weekly individual 50 minute psychotherapy sessions.
  Interventions: Behavioral: face-to-face individual therapy

INTERVENTIONS:
Behavioral: Therapist assisted online treatment — 7 weekly interactive online modules with 10-15 minute counselor consultation via video conference.
  Arms: Therapist assisted online treatment (TAO)
Behavioral: face-to-face individual therapy — weekly individual counseling as usual.
  Arms: face-to-face individual therapy

SUMMARY:
Therapist assisted, internet-based cognitive behavioral therapy (TAI-CBT) has been shown to be effective with patients who have Generalized Anxiety Disorder (GAD) in multiple studies from several countries, including: the United Kingdom, Australia, Sweden, and the Netherlands. Despite strong evidence of efficacy, TAI-CBT has not been offered in the USA. TAI-CBT could provide an effective alternative to face-to-face psychotherapy that would expand the availability and convenience of evidence- based treatment anywhere clinical availability is limited. The University of Florida (UF) has historically had greater demand for psychotherapy than the available supply of psychotherapy hours resulting in waiting lists for students needing to receive treatment for anxiety. Anxiety disorders interfere with memory and concentration thus impairing academic functioning. Students who must wait for treatment for 3-4 weeks are at risk for failing courses or dropping out of school. If TAI-CBT proved to be effective with UF students, providing it could increase the number of students who would receive effective and timely treatment. This project will create a 6-8 session therapist assisted on-line treatment for anxiety disorder. The investigators will offer TAI-CBT as an experimental treatment in summer and fall, 2013 comparing outcomes to face-to-face individual therapy, group therapy, and wait-list controls. The investigators hypothesize that students receiving TAI-CBT will have a reduction in anxiety symptoms comparable to face-to-face counseling and greater than wait list controls.

DETAILED DESCRIPTION:
Participation is restricted to currently enrolled students at the University of Florida who have paid the health fee, and who are seeking treatment for anxiety and the Counseling and Wellness Center. Students who meet criteria and agree to participate will select from two treatments, individual face-to-face or therapist assisted on-line treatment. Prior to each session of individual therapy, or on-line treatment participants will complete the Behavioral Health Measure-20 is a normal part of treatment at the CWC.

If a participant is assigned to the Therapist-assisted on-line (TAO) treatment he/she will be asked to complete a seven module on-line treatment. Each module includes interactive, educational materials and weekly assignments. Subjects may participate in an on-line discussion forum with other participants for each module. The forum will use only first names or a pseudonym to protect confidentiality. In addition, participants in the TAO treatment will receive a 10-20 minute video-conference weekly with a doctoral level therapist. Therapists will review assignments, answer questions, and help to apply the educational materials contained in the modules to the subjects life.

The video conference will be on Adobe Connect. This involves a free download for a computer, tablet, or smart phone. Medical records will be kept for ten years, per UF policy. Adobe connect is HIPAA and HITECH compliant. Research records will be de-identified and use an identifier number that cannot be connected to individual participants.

Only 2 arms were actually used, Face-to-face therapy and TAO treatment.

ELIGIBILITY:
Inclusion Criteria:

* students,
* mild to moderate anxiety,
* has appropriate computer equipment

Exclusion Criteria:

* Severe depression or anxiety,
* suicidal in past 12 months,
* not stable on medications for at least 30 days prior to beginning study treatments

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Behavioral Health Measure-20 (BHM-20) | The three measures will be administered weekly from initial enrollment in the study for 7 weeks and again at 6 month follow up. The first assessment of patients will begin May 7 and will continue through January, 2014.
  twenty item likert-type measure of distress, well-being, overall mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A Benton, Ph.D., Principal Investigator — University of Florida
Locations (1):
- Counseling and Wellness Center, University of Florida, Gainesville, Florida, United States